CLINICAL TRIAL: NCT01023152
Title: Effect of Remote Ischemic Preconditioning on Acute Kidney Injury in Patients Undergoing Heart Valve Replacement Surgery With Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Young Lan Kwak / Professor, Department of Anesthesiology and Pain Medicine, Severance Hospital
Model: Parallel | Purpose: Prevention
Other Study IDs: 4-2008-0423
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Heart Valve Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Automated cuff-inflator (Experimental)
  Interventions: Procedure: Automated cuff-inflator

INTERVENTIONS:
Procedure: Automated cuff-inflator — RIPC protocol consisted of three 10-min cycles of lower limb ischemia at an inflation pressure of 250 mmHg induced by an automated cuff-inflator placed on the upper leg with an intervening 10 min of reperfusion during which the cuff was deflated.

SUMMARY:
The purpose of this study is to study the effect of remote ischemic preconditioning on acute kidney injury in patients undergoing heart valve replacement surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
Hypothesis : RIPC using tourniquet might be a simple technique with the benefit to provide renal protection without disturbing operating procedure and prolongation of total operating time.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing complex valve surgery.

Exclusion Criteria:

* older than 80 years
* those with left main disease >50%, or hepatic or pulmonary disease
* active infective endocarditis
* left ventricular ejection fraction <30%
* myocardial infarction (MI) within 3 weeks
* pre-existing renal dysfunction (serum creatinine (Cr) level >1.4 mg/dl), and those with peripheral vascular disease affecting the lower limbs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)